CLINICAL TRIAL: NCT00049712
Title: A Phase I Study Of Medi 522 In Patients With Advanced Tumors
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Refractory Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000257810; P30CA014520 (NIH); WCCC-CO-01905; NCI-5497
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2015-07

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; intraocular lymphoma; primary central nervous system lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; small intestine lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult T-cell leukemia/lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; unspecified adult solid tumor, protocol specific; stage IV adult lymphoblastic lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage III adult T-cell leukemia/lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — etaracizumab

INTERVENTIONS:
Biological: etaracizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibody therapy in treating patients who have refractory advanced solid tumors or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of monoclonal antibody anti-alpha V beta 3 integrin (MEDI 522) in patients with refractory advanced solid tumors or lymphoma.
* Determine the safety and tolerability of this drug in these patients.
* Demonstrate significant binding of this drug to its molecular target in vivo in these patients.
* Determine the effects of this drug on angiogenesis in these patients.
* Determine antitumor activity of this drug by measuring tumor size and glucose uptake in these patients.
* Determine the pharmacokinetics of this drug in these patients.
* Determine a recommended phase II dose of this drug based on either the MTD or the optimal biologic response in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive monoclonal antibody anti-alpha V beta 3 integrin (Medi 522) IV over 30 minutes weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of Medi 522 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: Approximately 6-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor or lymphoma that is refractory to currently available standard therapies or for which there are no curative therapies
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* More than 12 weeks

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No prior bleeding disorder

Hepatic

* Bilirubin normal
* AST/ALT no greater than 2.5 times upper limit of normal
* INR/PTT normal

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation
* HIV negative
* T4 or thyroid stimulating hormone normal
* No thyroid disease
* No prior allergic reactions attributed to compounds of similar chemical or biologic composition to study drug (e.g., rituximab or immunoglobulin G)
* No ongoing or active infection
* No other uncontrolled concurrent illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered

Surgery

* More than 4 weeks since prior surgery

Other

* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies (commercial or investigational)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas McNeel, MD, PhD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States